CLINICAL TRIAL: NCT03119246
Title: Beta Testing of a New Assessment Protocol for Assessment of Complex Therapies in Huntington's Disease (HD)
Brief Title: Beta Testing of a New Assessment in Huntington's Disease (HD)
Acronym: CAPIT-HD Beta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: School of Biosciences - Cardiff University (Unknown); University Hospital of Wales (Other); National Reference Center for Huntington's disease Cognitive Neurology Unit (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Manchester Centre for Genomic Medicine - St. Mary's Hospital University of Manchester (Unknown); George-Huntington-Institut GmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P150201
Record Dates: First submitted 2016-08-25; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2016-08

CONDITIONS: Huntington Disease
Keywords: beta testing; assessment battery; HD
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HD patients (Experimental)
  Interventions: Other: CAPIT-HD beta
- Controls (Experimental)
  Interventions: Other: CAPIT-HD beta

INTERVENTIONS:
Other: CAPIT-HD beta — New assessment protocol for assessment of complex therapies in Huntington's disease for both groups

SUMMARY:
Huntington's disease (HD) is an inherited neurodegenerative disease for which there are no existing disease-modifying treatments.

Repair-HD is an EU FP7 consortium that aims to establish all the preclinical requirements for transplantation of stem cell-derived neurons in HD in order to replace those lost to the disease process. These requirements include the generation of new clinical assessments for detailed monitoring of patients with HD who have undergone cell replacement therapy.

This protocol describes the beta testing of a new clinical assessment battery: Core Assessment Protocol for Intrastriatal Transplantation in HD version 2 (CAPIT-HD beta / CAPIT-HD2). CAPIT-HD beta represents a substantial revision of a previous CAPIT-HD battery published over 20 years ago, which is in need of updating in order to accommodate knowledge from clinical transplant studies over this time and to take advantage of technological advances in patient assessment.

HD is a complex disorder in which there is relentless deterioration of motor, cognitive and behavioural functions, usually from mid-life onwards. The original CAPIT battery aimed to capture elements of change in all three domains, but was based predominantly on subjective semi-quantitative assessment tools that have poor inter-rater reliability. Moreover, a number of deficits, such as impairments in social cognition, were not recognised when the original CAPIT-HD battery was constructed, so we have developed novel assessments of these deficits, some of which are included in CAPIT-HD beta. The beta testing will take place in established HD clinical centres in Cardiff, Manchester, Paris, and Munster by teams of researchers who are experienced in leading clinic research in HD. Patients with early to moderate HD will be assessed at baseline, and at one and twelve months later, to assess the reliability and sensitivity of the CAPIT-HD beta battery. Arrangements for data storage and analysis are in place.

ELIGIBILITY:
1. Patients Inclusion criteria

   * Must be confirmed to carry the HD gene through genetic testing (CAG ≥ 36)
   * Must be 18 years or above
   * Stage I or II disease (TFC staging)

   Exclusion criteria
   * The inability to approve consent
   * Any comorbid condition that has the potential to confound the results of the study
2. Controls Inclusion criteria - Must be 18 years or above

Exclusion criteria

* The inability to approve consent
* Any comorbid condition that has the potential to confound the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
All dysfunction or disorder of huntington patient measured by means of a new battery assessments | 1 year
  The goal is to validate a battery of assessments for application in a wide range of complex therapies for Huntington's disease (HD)

SECONDARY OUTCOMES:
Difference on motor score between patient and healthy volontary measured by motor tests of the revised Core Assessment Protocol | 1 year
  The goal is to validate the discriminative ability of the revised Core Assessment Protocol for Intracranial transplantation in HD for the motor
Difference on cognitive score between patient and healthy volontary measured by cognitive tests of the revised Core Assessment Protocol | 1 year
  The goal is to validate the discriminative ability of the revised Core Assessment Protocol for Intracranial transplantation in HD for the cognitive
Difference on psychiatric score between patient and healthy volontary measured by psychiatric evaluation of the revised Core Assessment Protocol | 1 year
  The goal is to validate the discriminative ability of the revised Core Assessment Protocol for Intracranial transplantation in HD for the psychiatric
Difference on functional scale between patient and healthy volontary measured by functional evaluation of the revised Core Assessment Protocol | 1 year
  The goal is to validate the discriminative ability of the revised Core Assessment Protocol for Intracranial transplantation in HD for the functional domains of impairment in HD
Number of new assessment battery performed correctly | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Catherine BACHOUD-LEVI, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Anne ROSSER, MD, PhD, Principal Investigator — School of Biosciences - Cardiff University; David CRAUFURD, MD, PhD, Principal Investigator — Manchester Centre for Genomic Medicine - St. Mary's Hospital; Ralf REILMANN, MD, PhD, Principal Investigator — George-Huntington-Institut GmbH
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Derived] Chenain L, Riad R, Fraisse N, Jubin C, Morgado G, Youssov K, Lunven M, Bachoud-Levi AC. Graph methods to infer spatial disturbances: Application to Huntington's Disease's speech. Cortex. 2024 Jul;176:144-160. doi: 10.1016/j.cortex.2024.04.014. Epub 2024 May 17. PMID 38795650